CLINICAL TRIAL: NCT00770315
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Long-Term Safety of Ragweed (Ambrosia Artemisiifolia) Sublingual Tablet (SCH 39641) in Adult Subjects With a History of Ragweed-Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: Efficacy and Long-Term Safety of Ragweed (Ambrosia Artemisiifolia) Sublingual Tablet (SCH 39641) in Adults With a History of Ragweed-Induced Rhinoconjunctivitis With or Without Asthma (Study P05234)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05234; 3810249 (Other: Schering-Plough Study Number); 2008-003864-20 (EudraCT Number); MK-3641-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis, Allergic; Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SCH 39641 1.5 Amb a 1-U (Experimental): Participants receive Ambrosia artemisiifolia allergan extract (SCH 39641 1.5 Amb a 1-U) rapidly dissolving sublingual tablets, administered once daily for approximately 52 weeks
  Interventions: Biological: Ambrosia artemisiifolia allergen extract (Amb a 1-U)
- SCH 39641 6 Amb a 1-U (Experimental): Participants receive Ambrosia artemisiifolia allergan extract (SCH 39641 6 Amb a 1-U) rapidly dissolving sublingual tablets, administered once daily for approximately 52 weeks
  Interventions: Biological: Ambrosia artemisiifolia allergen extract (Amb a 1-U)
- SCH 39641 12 Amb a 1-U (Experimental): Participants receive Ambrosia artemisiifolia allergan extract (SCH 39641 12 Amb a 1-U) rapidly dissolving sublingual tablets, administered once daily for approximately 52 weeks
  Interventions: Biological: Ambrosia artemisiifolia allergen extract (Amb a 1-U)
- Placebo (Placebo Comparator): Participants receive matching placebo rapidly dissolving sublingual tablets, administered once daily for approximately 52 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ambrosia artemisiifolia allergen extract (Amb a 1-U) — Rapidly dissolving tablet administered sublingually once daily, at a dose of 1.5, 6 or 12 units.
  Other Names: SCH 39641; MK-3641
  Arms: SCH 39641 1.5 Amb a 1-U; SCH 39641 12 Amb a 1-U; SCH 39641 6 Amb a 1-U
Biological: Placebo — Placebo matching Ambrosia artemisiifolia allergen extract rapidly dissolving tablet, administered sublingually once daily
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ragweed sublingual tablet (SCH 39641/MK-3641/Amb a 1-U) compared with placebo in participants with ragweed-induced rhinoconjunctivitis over a one-year period. It is expected that ragweed allergic participants on one of the active arms of the trial will have decreased allergic rhinoconjunctivitis symptoms and require less allergy rescue medications during ragweed pollen season.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical history of significant ragweed-induced allergic rhinoconjunctivitis of at least 2 years duration, with or without asthma and have received treatment during the previous ragweed season (RS).
* Must have a positive skin prick test response to Ambrosia artemisiifolia at Screening Visit.
* Must be positive for specific immunoglobulin E (IgE) against Ambrosia artemisiifolia at Screening Visit.
* Must have an forced expiratory volume in one second (FEV1) of at least 70% of predicted at Screening Visit.
* Safety laboratory tests and vital signs conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor.
* Must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Female participants of childbearing potential must be using a medically acceptable and adequate form of birth control. These include: hormonal contraceptives as prescribed by a physician (oral, hormonal vaginal ring, hormonal implant or depot injectable); medically prescribed intra-uterine device; medically prescribed topically-applied transdermal contraceptive patch; double-barrier method (eg, condom in combination with a spermicide).
* Female participants of childbearing potential should be counseled in the appropriate use of birth control while in the study. Female participants who are not currently sexually active must and consent to use one of the above-mentioned methods if she becomes sexually active during the study.
* Female participants of childbearing potential must have a negative urine pregnancy test at Screening Visit. Women who have been surgically sterilized or at least 1 year postmenopausal are not considered to be of childbearing potential.

Exclusion Criteria:

* Clinical history of symptomatic seasonal allergic rhinitis and/or asthma having received regular medication, due to another during or potentially overlapping the RS.
* Clinical history of significant symptomatic perennial allergic rhinitis and/or asthma due to an allergen to which the participant is regularly exposed.
* Receipt of an immunosuppressive treatment within 3 months prior to the Screening Visit (except steroids for allergic and asthma symptoms).
* Clinical history of severe asthma.
* Asthma requiring medium or high dose inhaled corticosteroids (ICS).
* History of anaphylaxis with cardiorespiratory symptoms.
* History of chronic urticaria and angioedema.
* Clinical history of chronic sinusitis 2 years prior to the Screening Visit.
* Current severe atopic dermatitis.
* Breast-feeding, pregnancy, or intending to become pregnant.
* Had previous treatment by immunotherapy with ragweed allergen or any other allergen 5 years prior to Screening Visit.
* History of allergy, hypersensitivity or intolerance to the ingredients of the investigational medicinal products (except for Ambrosia artemisiifolia), rescue medications, or self-injectable epinephrine.
* Any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.
* Use of any investigational drugs within 30 days of Screening Visit.
* Participation in any other clinical study.
* Being a family member of the study staff.
* Inability to meet medication washout requirements.
* Unlikely to be able to complete the trial, or likely to travel for an extended time during the RS.
* Clinically significant abnormal vital sign or lab value.
* Participation in this same study at another site.
* Randomized into this study more than once.
* Inability to or will not comply with the use of self-injectable epinephrine.
* Greater risk of developing adverse reactions after epinephrine administration.
* History of self-injectable epinephrine use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 784 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

REFERENCES:
- [Result] Creticos PS, Maloney J, Bernstein DI, Casale T, Kaur A, Fisher R, Liu N, Murphy K, Nekam K, Nolte H. Randomized controlled trial of a ragweed allergy immunotherapy tablet in North American and European adults. J Allergy Clin Immunol. 2013 May;131(5):1342-9.e6. doi: 10.1016/j.jaci.2013.03.019. PMID 23622121
- [Derived] Christensen LH, Ipsen H, Nolte H, Maloney J, Nelson HS, Weber R, Lund K. Short ragweeds is highly cross-reactive with other ragweeds. Ann Allergy Asthma Immunol. 2015 Dec;115(6):490-495.e1. doi: 10.1016/j.anai.2015.09.016. Epub 2015 Oct 21. PMID 26507708
- [Derived] Kim H, Waserman S, Hebert J, Blaiss M, Nelson H, Creticos P, Kaur A, Maloney J, Li Z, Nolte H. Efficacy and safety of ragweed sublingual immunotherapy in Canadian patients with allergic rhinoconjunctivitis. Allergy Asthma Clin Immunol. 2014 Nov 10;10(1):55. doi: 10.1186/1710-1492-10-55. eCollection 2014. PMID 25788949
- [Derived] Nolte H, Amar N, Bernstein DI, Lanier BQ, Creticos P, Berman G, Kaur A, Hebert J, Maloney J. Safety and tolerability of a short ragweed sublingual immunotherapy tablet. Ann Allergy Asthma Immunol. 2014 Jul;113(1):93-100.e3. doi: 10.1016/j.anai.2014.04.018. Epub 2014 May 14. PMID 24836393

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants receive placebo matching Ambrosia artemisiifolia allergan extract rapidly dissolving sublingual tablets, administered once daily for approximately 52 weeks
Period: Overall Study
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Started | 197 | 195 | 194 | 198
Completed | 157 | 152 | 137 | 160
Not Completed | 40 | 43 | 57 | 38
Not completed — Adverse Event | 11 | 17 | 16 | 6
Not completed — Lost to Follow-up | 9 | 5 | 10 | 3
Not completed — Withdrawal by Subject | 13 | 17 | 24 | 20
Not completed — Noncompliance with Protocol | 7 | 4 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo | Total
Number analyzed (Participants) | 197 | 195 | 194 | 198 | 784
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.83) | 36.9 (8.80) | 35.6 (8.75) | 36.7 (8.54) | 36.4 (8.73)
Gender [Count of Participants; unit: Participants]
  Female | 110 | 103 | 91 | 96 | 400
  Male | 87 | 92 | 103 | 102 | 384

OUTCOME MEASURES:

1. Primary Outcome: Combined (Sum of) Rhinoconjunctivitis Daily Symptom Score (DSS) and Daily Medication Score (DMS) Averaged Over the Peak Ragweed Season (RS)
Description: The total combined score is a composite endpoint that combines the rhinoconjuntivitis DSS and the rhinoconjunctivitis DMS. The rhinoconjunctivitis DSS consisted of a total of 6 symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes and watery eyes) that were measured on a scale of 0 to 3 (0=no symptoms, 3=severe symptoms; score range: 0-18), with a lower score indicating less rhinoconjunctivitis symptoms. Rhinoconjunctivitis DMS was based on use of specific study-provided rescue medication, with different rescue medications being assigned different scores/dose unit (score range: 0-36), with a lower score indicating less rhinconjunctivitis medication use. The sum of the rhinoconjunctivitis DSS+DMS could range from 0 to 54, with a lower score indicating less rhinoconjuntivitis symptoms and medication use. Raw means were converted to adjusted means using an ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: The Full Analysis Set (FAS) population consisted of all randomized participants who took at least one dose of study medication and had at least one post-randomization efficacy measurement.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 169 | 167 | 152 | 169
score on a scale | 7.70 (0.517) [-1.98 to 0.45] | 6.88 (0.526) [-2.80 to -0.36] | 6.41 (0.534) [-3.30 to -0.79] | 8.46 (0.535) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 1.5 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.2192, ANOVA; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-1.98 to 0.45] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0113, ANOVA; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-2.80 to -0.36] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 3: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0015, ANOVA; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-3.30 to -0.79] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

2. Secondary Outcome: Average Combined Rhinoconjunctivitis DSS and DMS Over the Entire RS
Description: as for outcome 1
Time Frame: Approximately 5 weeks
Population: The FAS population consisted of all randomized participants who took at least one dose of study medication and had at least one post-randomization efficacy measurement.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 171 | 172 | 158 | 174
score on a scale | 6.22 (0.432) [-1.88 to 0.13] | 5.81 (0.433) [-2.29 to -0.28] | 5.18 (0.439) [-2.95 to -0.88] | 7.09 (0.441) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 1.5 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0878, ANOVA; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.88 to 0.13] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0125, ANOVA; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.29 to -0.28] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 3: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0003, ANOVA; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-2.95 to -0.88] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

3. Secondary Outcome: Average Rhinoconjunctivitis DSS for the Peak RS
Description: The rhinoconjunctivitis DSS consisted of a total of 6 symptoms (runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy eyes and watery eyes) that were measured on a scale of 0 to 3 (0=no symptoms, 3=severe symptoms; score range: 0-18), with a lower score indicating less rhinoconjunctivitis symptoms. Raw means were converted to adjusted means using an ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 169 | 167 | 152 | 169
score on a scale | 5.11 (0.301) [-0.96 to 0.45] | 4.87 (0.306) [-1.21 to 0.21] | 4.43 (0.311) [-1.67 to -0.21] | 5.37 (0.311) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 1.5 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.4781, ANOVA; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.96 to 0.45] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.1695, ANOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.21 to 0.21] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 3: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0118, ANOVA; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.67 to -0.21] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

4. Secondary Outcome: Average Rhinoconjunctivitis DSS for the Entire RS
Description: as for outcome 3
Time Frame: Approximately 5 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 171 | 172 | 158 | 174
score on a scale | 4.24 (0.255) [-0.93 to 0.25] | 4.19 (0.256) [-0.99 to 0.20] | 3.62 (0.259) [-1.57 to -0.35] | 4.58 (0.261) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 1.5 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.2622, ANOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.93 to 0.25] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.1914, ANOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.99 to 0.20] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 3: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0021, ANOVA; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.57 to -0.35] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

5. Secondary Outcome: Average Rhinoconjunctivitis DMS for the Peak RS
Description: Rhinoconjunctivitis DMS was based on participant use of specific study-provided rescue medication, with different rescue medications being assigned different scores/dose unit (score range: 0-36), with a lower score indicating less rhinconjunctivitis medication use. Raw means were converted to adjusted means using an ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects.
Time Frame: The 15-day period during the ragweed season with the highest moving pollen average
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Number analyzed (Participants) | 169 | 167 | 152 | 169
score on a scale | 2.58 (0.322) [-1.26 to 0.25] | 2.01 (0.328) [-1.84 to -0.32] | 1.99 (0.333) [-1.89 to -0.32] | 3.09 (0.333) [NA to NA]
Statistical Analysis 1: Comparison: SCH 39641 1.5 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.1900, ANOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.26 to 0.25] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 2: Comparison: SCH 39641 6 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0053, ANOVA; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-1.84 to -0.32] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects
Statistical Analysis 3: Comparison: SCH 39641 12 Amb a 1-U vs Placebo; Test type: Superiority or Other; p = 0.0058, ANOVA; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-1.89 to -0.32] — ANOVA model with baseline asthmatic condition, pollen region and treatment group as fixed effects

ADVERSE EVENTS:
Time Frame: Up to 53 weeks
Description: The population consisted of all randomized participants who took at least one dose of study medication.
Arm/Group | SCH 39641 1.5 Amb a 1-U | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Placebo
Serious Adverse Events (participants affected / at risk) | 5/196 | 4/195 | 4/194 | 1/198
Other Adverse Events (participants affected / at risk) | 105/196 | 108/195 | 125/194 | 78/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 39641 1.5 Amb a 1-U (N=196) | SCH 39641 6 Amb a 1-U (N=195) | SCH 39641 12 Amb a 1-U (N=194) | Placebo (N=198)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 39641 1.5 Amb a 1-U (N=196) | SCH 39641 6 Amb a 1-U (N=195) | SCH 39641 12 Amb a 1-U (N=194) | Placebo (N=198)
Ear pruritus (Ear and labyrinth disorders) | 14 (15) | 27 (30) | 25 (26) | 2 (2)
Oral pruritus (Gastrointestinal disorders) | 11 (12) | 29 (37) | 16 (17) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 10 (11) | 15 (18) | 9 (14) | 5 (9)
Swollen tongue (Gastrointestinal disorders) | 11 (11) | 12 (14) | 15 (16) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 8 (8) | 15 (16) | 12 (14) | 0 (0)
Tongue pruritus (Gastrointestinal disorders) | 13 (14) | 19 (26) | 18 (21) | 3 (3)
Bronchitis (Infections and infestations) | 5 (7) | 6 (6) | 8 (8) | 12 (14)
Nasopharyngitis (Infections and infestations) | 31 (40) | 28 (35) | 33 (42) | 35 (45)
Sinusitis (Infections and infestations) | 12 (13) | 9 (10) | 8 (9) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 18 (22) | 9 (12) | 9 (11)
Headache (Nervous system disorders) | 15 (33) | 12 (17) | 18 (49) | 20 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 10 (10) | 12 (14) | 6 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 5 (5) | 9 (10) | 4 (4)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 6 (7) | 8 (10) | 4 (8)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 42 (46) | 41 (45) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.